CLINICAL TRIAL: NCT03815383
Title: A Phase Ⅰ Study Evaluating Safety and Efficacy of C-CAR088 Treatment in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of BCMA-directed CAR-T Cells Treatment in Subjects With r/r Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0203-008
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2018-12

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR088 (Experimental): Lymphocytes will be transduced with lentiviral vector containing CAR-BCMA gene
  Interventions: Biological: C-CAR088

INTERVENTIONS:
Biological: C-CAR088 — Autologous BCMA-directed CAR-T cells by a single infusion intravenously will be given in escalating doses.
  Other Names: CBM.BCMA Chimeric Antigen Receptor T cell

SUMMARY:
This is a single-center, non-randomized and dose-escalation study to evaluate the safety and efficacy of C-CAR088 in relapsed or refractory multiple myeloma patient.

DETAILED DESCRIPTION:
The study will include the following sequential phases: Screening, Pre- Treatment (Cell Product Preparation, Lymphodepleting Chemotherapy), C-CAR088 infusion and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate in this study and signed informed consent.
2. Age 18-75 years old, male or female.
3. Meet the internationally accepted Criteria for the diagnosis of multiple myeloma (IMWG diagnostic criteria 2014).
4. Patients with relapsed or refractory multiple myeloma.
5. Subjects have one or more measurable multiple myeloma lesion, must include one of the following conditions:

   * Serum M protein≥1 g/dl(10g/L)
   * Urine M protein≥200 mg/24h
   * Serum free light chain(sFLC): κ/λ ratio abnormal and ≥10 mg/dl
6. Bone marrow sample is confirmed as BCMA-positive by flow cytometry or pathological examination.
7. At least 2 weeks from monoclonal antibody therapy prior to CAR T cell therapy.
8. ECOG scores 0 - 1.
9. Normal cardiac diastolic function, left ventricular ejection fraction (LVEF) ≥ 50% (detected by echocardiography), no serious arrhythmia.
10. No active pulmonary infections, normal pulmonary function and oxygen saturation ≥ 92% on room air.
11. No contraindications of leukapheresis.
12. Expected survival > 12 weeks.
13. Female subjects in childbearing age, their serum or urine pregnancy test must be negative,until 7 days before cell therapy and all subjects must agree to take effective contraceptive measures during the trial.

Exclusion Criteria:

1. Have a history of allergy to cellular products.
2. Any kind of these laboratory testing: including but not limited to,serum total bilirubin≧1.5mg/dl, serum ALT, AST≧2.5×ULN, serum creatinine≧2.0mg/dl, Hb (hemoglobin)<80g/L, neutrophils<1000/mm^3, platelets≦50000/mm^3 or platelet count maintained by transfusion.
3. Subjects with the clinically significant cardiovascular diseases.
4. A history of craniocerebral trauma, consciousness disorder, epilepsy, severe cerebral ischemia or hemorrhagic disease.
5. Use any anticoagulant (except aspirin).
6. Patients requiring urgent treatment due to tumor progression or spinal cord compression.
7. Patients with active CNS involvement or clinical syndrome of MM meningeal involvement.
8. After allogeneic hematopoietic stem cell transplantation.
9. Plasma cell leukemia.
10. Subjects with any autoimmune disease or any immune deficiency disease or other disease in need of immunosuppressive therapy.
11. Uncontrolled active infection.
12. Prior treatment with CAR T therapy or any other genetically modified T cell therapy.
13. Live vaccine inoculation within four weeks before enrollment.
14. Hepatitis B or hepatitis C virus infection (including carriers), syphilis, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV-infected persons.
15. Have a history of alcoholism, drug addiction and mental illness.
16. Participated in any other clinical trial within one month.
17. The investigators believe that there are other circumstances that are not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Safety:TEAEs | 30 days
  The incidence of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
ORR | 12 months
  Overall response rate
PFS | 6 months, 12 months
  Progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Qu X, An G, Sui W, Wang T, Zhang X, Yang J, Zhang Y, Zhang L, Zhu D, Huang J, Zhu S, Yao X, Li J, Zheng C, Zhu K, Wei Y, Lv X, Lan L, Yao Y, Zhou D, Lu P, Qiu L, Li J. Phase 1 study of C-CAR088, a novel humanized anti-BCMA CAR T-cell therapy in relapsed/refractory multiple myeloma. J Immunother Cancer. 2022 Sep;10(9):e005145. doi: 10.1136/jitc-2022-005145. PMID 36100310